CLINICAL TRIAL: NCT04336189
Title: Optimal Chemopreventive Regimens to Prevent Malaria and Improve Birth Outcomes in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grant Dorsey, M.D, Ph.D. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Infectious Diseases Research Collaboration, Uganda (Other)
Responsible Party: Sponsor-Investigator, Grant Dorsey, M.D, Ph.D., Principle Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: DPSP
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-06

CONDITIONS: Malaria
Keywords: dihydroartemisinin-piperaquine; sulfadoxine-pyrimethamine; IPTp; reproductive tract infection; microbiome; drug resistance
MeSH Terms: conditions — Malaria; Reproductive Tract Infections | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two drugs on day 1 (SP and placebo or DP and placebo or SP and DP) followed by one drug on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP. A randomization list will be computer generated by a member of the project who will not be directly involved in the conduct of the study. The randomization list will include consecutive treatment numbers with corresponding random treatment assignments. Randomized codes will correspond to the 3 treatment arms using permuted variable sized blocks of 6 and 9.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SP + DP placebo every 4 weeks (Active Comparator)
  Interventions: Drug: Sulfadoxine-pyrimethamine (SP)
- DP + SP placebo every 4 weeks (Active Comparator)
  Interventions: Drug: Dihydroartemisinin-piperaquine (DP)
- SP + DP given every 4 weeks (Active Comparator)
  Interventions: Drug: Sulfadoxine-pyrimethamine (SP); Drug: Dihydroartemisinin-piperaquine (DP)

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine (SP) — SP (Kamsidar) will be supplied by Kampala Pharmaceutical Industries (KPI), Uganda. SP will be given as a single dose consisting of 3 full strength tablets.
  Other Names: Kamsidar
  Arms: SP + DP given every 4 weeks; SP + DP placebo every 4 weeks
Drug: Dihydroartemisinin-piperaquine (DP) — DP (Duo-Cotecxin) will be supplied by Holley-Cotec, Beijing, China. DP will consist of 3 full strength tablets given once a day for 3 consecutive days.
  Other Names: Duo-Cotecxin
  Arms: DP + SP placebo every 4 weeks; SP + DP given every 4 weeks

SUMMARY:
This trial tests the hypothesis that intermittent preventive treatment in pregnancy (IPTp) with sulfadoxine-pyrimethamine (SP) + dihydroartemisin-piperaquine (DP) will significantly reduce the risk of adverse birth outcomes compared to IPTp with SP alone or DP alone. This double-blinded randomized controlled phase III trial of 2757 HIV uninfected pregnant women enrolled at 12-20 weeks gestation will be randomized in equal proportions to one of three IPTp treatment arms: 1) SP given every 4 weeks, or 2) DP given every 4 weeks, or 3) SP+DP given every 4 weeks. SP or DP placebos will be used to ensure adequate blinding is achieved in the study and follow-up will end 28 days after giving birth.

DETAILED DESCRIPTION:
Malaria in pregnancy remains a major challenge in Africa, where approximately 50 million women are at risk for P. falciparum infection during pregnancy each year. Among pregnant women living in malaria endemic areas symptomatic disease is uncommon, but infection with malaria parasites is associated with maternal anemia and adverse birth outcomes including abortions, stillbirth, preterm birth, low birth weight (LBW), and infant mortality. The World Health Organization (WHO) recommends the use of long-lasting insecticidal nets (LLINs) and intermittent preventive treatment with sulfadoxine-pyrimethamine (IPTp-SP) for the prevention of malaria in pregnancy in endemic areas of Africa. However, there is concern for diminishing efficacy of these interventions due to the spread of vector resistance to the pyrethroid insecticides used in LLINs and parasite resistance to SP. Thus, there is an urgent need for new strategies for the prevention of malaria in pregnancy and improving birth outcomes. Artemisinin-based combination therapies (ACTs) are now the standard treatment for malaria in Africa. Dihydroartemisin-piperaquine (DP) is a fixed-dose ACT and an attractive alternative to SP for IPTp. DP is highly efficacious, and the long half-life of piperaquine provides at least 4 weeks of post-treatment prophylaxis. Recent randomized controlled trials showed that, compared to IPTp with SP, IPTp with DP dramatically reduced risks of malaria-specific outcomes but there were minimal differences between the SP and DP groups in risks of adverse birth outcomes. The key question for this study is why IPTp with either SP or DP is associated with similar risks of adverse birth outcomes despite the far superior antimalarial activity of DP. The likely explanation is that SP, a broad-spectrum antibiotic, protects against non-malarial causes of LBW and preterm birth. The central hypothesis is that SP improves birth outcomes independent of its antimalarial activity and that IPTp with a combination of SP+DP will offer antimalarial and non-antimalarial benefits, thus providing superior prevention of adverse birth outcomes compared to either drug used alone. To test this hypothesis, a double-blinded randomized clinical trial will conducted in a rural area of Uganda with very high malaria transmission intensity, where there is already an established infrastructure for clinical research. Specific aims will be (1) to compare the risk of adverse birth outcomes among pregnant women randomized to receive monthly IPTp with SP vs. DP vs. SP+DP, (2) To compare safety and tolerability of IPTp regimens among pregnant women randomized to receive monthly IPTp with SP vs. DP vs. SP+DP, and (3) to compare risks of malaria-specific and non-malarial outcomes among pregnant women randomized to receive monthly IPTp with SP vs. DP vs. SP+DP. This study will be the first to evaluate the efficacy and safety of a novel combination of well-studied drugs for improving birth outcomes and findings may well have important policy implications, with a change in standard practice for millions of pregnant women in Africa.

ELIGIBILITY:
Inclusion Criteria:

1. Viable singleton pregnancy confirmed by ultrasound
2. Estimated gestational age between 12-20 weeks
3. Confirmed to be HIV- uninfected by rapid test
4. 16 years of age or older
5. Residency within Busia District of Uganda
6. Provision of informed consent
7. Agreement to come to the study clinic for any febrile episode or other illness and avoid medications given outside the study protocol
8. Willing to deliver in the hospital

Exclusion Criteria:

1. History of serious adverse event to SP or DP
2. Active medical problem requiring inpatient evaluation at the time of screening
3. Intention of moving outside of Busia District Uganda
4. Chronic medical condition requiring frequent medical attention
5. Prior chemopreventive therapy or any other antimalarial therapy during this pregnancy
6. Early or active labor (documented by cervical change with uterine contractions)
7. Multiple pregnancies (i.e. twins/triplets)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 2757 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco; Phil Rosenthal, MD, Principal Investigator — University of California, San Francisco; Moses Kamya, MBChB, MMed, PhD, Principal Investigator — Makerere University; Infectious Diseases Research Collaboration; Abel Kakuru, MBChB, PhD, Study Director — Infectious Diseases Research Collaboration
Locations (1):
- Infectious Diseases Research Collaboration Clinic - Masafu Hospital, Masafu, Busia, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kakuru A, Kizza J, Aguti M, Adrama H, Ategeka J, Olwoch P, Nakalembe M, Nankabirwa JI, Opira B, Ozarslan N, Ranjit A, Dela Cruz E, Clark TD, Roh ME, Gaw SL, Jagannathan P, Rosenthal PJ, Kamya MR, Dorsey G. Dihydroartemisinin-piperaquine plus sulfadoxine-pyrimethamine versus either drug alone for intermittent preventive treatment of malaria in pregnancy: A double-blind, randomized, controlled phase 3 trial from Uganda. PLoS Med. 2025 Sep 18;22(9):e1004582. doi: 10.1371/journal.pmed.1004582. eCollection 2025 Sep. PMID 40966190

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Started | 918 | 920 | 919
Completed | 842 | 846 | 850
Not Completed | 76 | 74 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks | Total
Number analyzed (Participants) | 918 | 920 | 919 | 2757
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (6.2) | 24.7 (6.3) | 24.2 (6.0) | 24.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 918 | 920 | 919 | 2757
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 918 | 920 | 919 | 2757
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 918 | 920 | 919 | 2757
Gestational age [Mean (Standard Deviation); unit: weeks] | 15.8 (2.6) | 15.7 (2.5) | 16.0 (2.6) | 15.8 (2.6)
Gestational age categories [Count of Participants; unit: Participants]
  12-16 weeks | 522 | 530 | 481 | 1533
  >16 weeks | 396 | 390 | 438 | 1224
Gravidity [Count of Participants; unit: Participants]
  Primigravidae | 230 | 234 | 262 | 726
  Multigravidae | 688 | 686 | 657 | 2031
Bednet ownership [Count of Participants; unit: Participants]
  None | 423 | 434 | 415 | 1272
  Untreated net | 43 | 40 | 42 | 125
  Long-lasting insecticide-treated net | 452 | 446 | 462 | 1360
Household wealth index [Count of Participants; unit: Participants] — Population: Data not collected from 29 participants
  Participants
    number analyzed (Participants) | 908 | 909 | 911 | 2728
    Lowest tertile | 308 | 294 | 295 | 897
    Middle tertile | 293 | 319 | 309 | 921
    Highest tertile | 307 | 296 | 307 | 910
Highest level of education [Count of Participants; unit: Participants]
  None | 44 | 31 | 36 | 111
  Primary school | 592 | 593 | 600 | 1785
  Secondary school | 263 | 276 | 264 | 803
  Higher | 19 | 20 | 19 | 58
Weight in kg [Mean (Standard Deviation); unit: kg] | 57.3 (9.4) | 57.6 (9.8) | 57.1 (8.9) | 57.4 (9.4)
Height in cm [Mean (Standard Deviation); unit: cm] | 159 (6) | 159 (7) | 159 (6) | 159 (6)
Maternal MUAC [Mean (Standard Deviation); unit: cm] | 26 (4) | 26 (3) | 26 (3) | 26 (3)
Mean hemoglobin [Mean (Standard Deviation); unit: g/dL] | 11.6 (1.3) | 11.7 (1.3) | 11.5 (1.4) | 11.6 (1.4)
Prevalence of dhfr/dhps quintuple mutant markers of antifolate resistance [Number; unit: participants] — Population: Randomly subset of 200 participant samples with parasite density >100/microliter
  participants
    dhfr/dhps quintuple mutant: number analyzed (Participants) | 72 | 65 | 63 | 200
    dhfr/dhps quintuple mutant | 72 | 64 | 62 | 198
    dhfr l164L: number analyzed (Participants) | 72 | 65 | 63 | 200
    dhfr l164L | 14 | 19 | 8 | 41
    dhps A581G: number analyzed (Participants) | 72 | 65 | 63 | 200
    dhps A581G | 1 | 2 | 1 | 4
Detection of malaria parasites by microscopy or qPCR [Count of Participants; unit: Participants] | 634 | 637 | 657 | 1928

OUTCOME MEASURES:

1. Primary Outcome: Risk of Having a Composite Adverse Birth Outcome
Description: Composite adverse birth outcome defined as the occurrence of any of the following:
  * Spontaneous abortion: Fetal loss at < 28 weeks gestational age
  * Stillbirth: Infant born deceased at > 28 weeks gestational age
  * Low Birth Weight (LBW): Live birth with birth weight < 2500 gm
  * Preterm birth: Live birth at < 37 weeks gestational age
  * Small-for-gestational age (SGA): Live birth with weight-for-gestational age < 10th percentile of reference population
  * Neonatal death: Live birth with neonatal death within the first 28 days of life
Time Frame: Time from first dose of study drugs up to 28 days postpartum, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 842 | 846 | 850
Participants | 222 | 261 | 255

2. Primary Outcome: Incidence of Serious Adverse Events (SAE) Per Time at Risk
Description: SAEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: Time from first dose of study drugs up to 28 days postpartum, an average of 6 months
Measure: Number; unit: Events per person-years
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-years | 0.06 | 0.06 | 0.06

3. Primary Outcome: Incidence of Any Grade 3 or 4 or Serious Adverse Events Per Time at Risk
Description: Grade 3 and 4 AEs or SAEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: Time from first dose of study drugs up to 28 days postpartum, an average of 6 months
Measure: Number; unit: Events per person-year
Units Other Than Participants: Person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (Person years) | 432 | 434 | 433
Events per person-year | 0.23 | 0.19 | 0.21

4. Secondary Outcome: Number of Participants With Spontaneous Abortion
Description: Spontaneous abortion defined as fetal loss at < 28 weeks gestational age
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 842 | 846 | 850
Participants | 12 | 16 | 13

5. Secondary Outcome: Incidence of Anemia Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: Day study drugs are first given until when study participants reach 28 days postpartum or early study termination, an average of 6 months
Measure: Number; unit: Events per person-years
Units Other Than Participants: Person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (Person years) | 432 | 434 | 433
Events per person-years | 53 | 28 | 44

6. Secondary Outcome: Incidence of Grade 3-4 AEs Possibly Related to Study Drugs
Description: Grade 3-4 AEs possibly or definitely related to study drug defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-years
Units Other Than Participants: Person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (Person years) | 432 | 434 | 433
Events per person-years | 50 | 29 | 41

7. Secondary Outcome: Risk of Placental Malaria
Description: Detection of malaria parasites or pigment by histopathology
Time Frame: At the time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 776 | 795 | 784
Participants | 472 | 324 | 393

8. Secondary Outcome: Incidence of Malaria During Pregnancy
Description: Episodes of symptomatic malaria (incidence per person year at risk following initiation of study drugs)
Time Frame: Day study drugs first given until delivery, an average of 6 months
Measure: Number; unit: Events per person-years
Units Other Than Participants: Person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (Person years) | 367 | 369 | 367
Events per person-years | 1.15 | 0.02 | 0.04

9. Secondary Outcome: Microscopic Parasitemia During Pregnancy
Description: Proportion of routine samples with asexual parasites detected by microscopy
Time Frame: Day study drugs first given until delivery, an average of 6 months
Measure: Number; unit: Routine visits with parasitemia
Units Other Than Participants: Routine visits
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (Routine visits) | 4350 | 4348 | 4354
Routine visits with parasitemia | 771 | 25 | 60

10. Secondary Outcome: Prevalence of Anemia During Pregnancy
Description: Proportion of routine hemoglobin measurements < 11 g/dL
Time Frame: Day study drugs are first given until delivery
Measure: Number; unit: Routine visits with anemia
Units Other Than Participants: Routine visits
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (Routine visits) | 2232 | 2252 | 2229
Routine visits with anemia | 965 | 827 | 880

11. Secondary Outcome: Stillbirth
Description: Stillbirth defined as infant born deceased at > 28 weeks gestational age
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 830 | 830 | 837
Participants | 15 | 16 | 7

12. Secondary Outcome: Low Birth Rate
Description: Low birth weight defined as live birth with birth weight < 2500 gm
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 815 | 812 | 830
Participants | 47 | 59 | 71

13. Secondary Outcome: Preterm Delivery
Description: Preterm delivery defined as live birth at < 37 weeks gestational age
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 815 | 814 | 830
Participants | 48 | 25 | 44

14. Secondary Outcome: Small-for-gestational Age
Description: Small-for-gestational age defined as live birth with weight-for-gestational age < 10th percentile of reference population
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 815 | 812 | 830
Participants | 152 | 206 | 194

15. Secondary Outcome: Neonatal Death
Description: Neonatal death defined as live birth with neonatal death within the first 28 days of life
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 815 | 814 | 830
Participants | 4 | 5 | 12

16. Secondary Outcome: Microscopic or Sub-microscopic Parasitemia During Pregnancy
Description: Proportion of routine samples with asexual parasites detected by microscopy or qPCR
Time Frame: Day study drugs first given until delivery, an average of 6 months
Measure: Number; unit: routine visits with parasitemia
Units Other Than Participants: routine visits
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (routine visits) | 4350 | 4348 | 4354
routine visits with parasitemia | 2099 | 551 | 60

17. Secondary Outcome: Prevalence of Severe Anemia During Pregnancy
Description: Proportion of routine hemoglobin measurements < 8 g/dL
Time Frame: Day study drugs are first given until delivery, an average of 6 months
Measure: Number; unit: Routine visits with severe anemia
Units Other Than Participants: Routine visits
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 918 | 902 | 908
Number analyzed (Routine visits) | 2232 | 2252 | 2229
Routine visits with severe anemia | 29 | 9 | 12

18. Secondary Outcome: Incidence of Stillbirth Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-year
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-year | 15 | 16 | 7

19. Secondary Outcome: Incidence of Congenital Anomaly Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-year
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-year | 4 | 13 | 10

20. Secondary Outcome: Incidence of Neutropenia Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-year
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-year | 5 | 10 | 7

21. Secondary Outcome: Incidence of Proteinuria Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-years
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-years | 3 | 4 | 8

22. Secondary Outcome: Incidence of Thrombocytopenia Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-years
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-years | 7 | 1 | 2

23. Secondary Outcome: Incidence of Postpartum Hemorrhage Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-years
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-years | 2 | 3 | 2

24. Secondary Outcome: Incidence of Pre-eclampsia Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-years
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-years | 3 | 0 | 2

25. Secondary Outcome: Incidence of Preterm Birth <28 Gestational Age Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-years
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-years | 0 | 0 | 3

26. Secondary Outcome: Incidence of Elevated Temperature Adverse Event Per Time at Risk
Description: Grade 3-4 AEs as defined by the July 2017 NIH DAIDS Toxicity Tables
Time Frame: as for outcome 5
Measure: Number; unit: Events per person-year
Units Other Than Participants: person years
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
Number analyzed (Participants) | 896 | 902 | 908
Number analyzed (person years) | 432 | 434 | 433
Events per person-year | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day study drugs are first given until when study participants reach 28 days postpartum or early study termination, an average of 6 months
Description: Division of AIDS (DAIDS) Table for grading the severity of adult and pediatric adverse events, version 2017
Arm/Group | SP + DP placebo every 4 weeks | DP + SP placebo every 4 weeks | SP + DP given every 4 weeks
All-Cause Mortality (participants affected / at risk) | 1/896 | 2/902 | 0/908
Serious Adverse Events (participants affected / at risk) | 25/896 | 26/902 | 27/908
Other Adverse Events (participants affected / at risk) | 896/896 | 902/902 | 908/908
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP + DP placebo every 4 weeks (N=896) | DP + SP placebo every 4 weeks (N=902) | SP + DP given every 4 weeks (N=908)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 2 (2) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 4 (4)
Post-partum hemmorrha (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 2 (2)
Septicemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Abruptio placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Congenital anomoly (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 13 (13) | 10 (10)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 2 (2)
Transverse myelitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Puerperal sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Deep laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP + DP placebo every 4 weeks (N=896) | DP + SP placebo every 4 weeks (N=902) | SP + DP given every 4 weeks (N=908)
Abdominal pain (Gastrointestinal disorders) | 620 (1532) | 621 (1431) | 584 (1364)
Cough (Respiratory, thoracic and mediastinal disorders) | 526 (1064) | 540 (1130) | 527 (1004)
Headache (Nervous system disorders) | 510 (947) | 477 (865) | 436 (769)
Dysuria (Renal and urinary disorders) | 267 (379) | 25 (324) | 240 (324)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 155 (189) | 138 (164) | 141 (167)
Diarrhea (Gastrointestinal disorders) | 136 (174) | 123 (143) | 114 (140)
Fatigue (General disorders) | 82 (101) | 62 (79) | 49 (56)
Chills (General disorders) | 67 (67) | 63 (90) | 55 (66)
Epigastric pain (Gastrointestinal disorders) | 56 (83) | 72 (79) | 60 (62)
Anemia (Blood and lymphatic system disorders) | 45 (45) | 26 (26) | 38 (38)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 16 (16) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (3) | 4 (4) | 8 (8)
Thrombocytopenia (Renal and urinary disorders) | 7 (7) | 1 (1) | 2 (2)
Preterm birth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3)
Elevated temperature (General disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04336189/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04336189/SAP_001.pdf